CLINICAL TRIAL: NCT00344123
Title: Pharmacokinetic Evaluation of Single-dose Rosuvastatin 10 mg When Co-administered With Steady-state Tipranavir 500 mg/Ritonavir 200 mg TPV/r) B.I.D. in Healthy Adult Volunteers
Brief Title: Pharmacokinetic (PK) Study of Single-dose Rosuvastatin and Tipranavir/Ritonavir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00003633
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tipranavir/ritonavir (Other): On Day 1, subjects will receive a single 10 mg dose of rosuvastatin.
  Beginning on Day 3, subjects will receive a combination of TPV 500mg/RTV 200 mg twice daily for 11 days (Days 3-13).
  On Day 12, subjects will receive a single 10 mg dose of rosuvastatin co-administered with TPV/r.
  Interventions: Drug: Tipranavir/Ritonavir; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Tipranavir/Ritonavir — On Day 1, subjects will receive a single 10 mg dose of rosuvastatin. Beginning on Day 3, subjects will receive a combination of TPV 500mg/RTV 200 mg twice daily for 11 days (Days 3-13).
  On Day 12, subjects will receive a single 10 mg dose of rosuvastatin co-administered with TPV/r.
  Other Names: Aptivus
Drug: Rosuvastatin — On Day 1, subjects will receive a single 10 mg dose of rosuvastatin. Beginning on Day 3, subjects will receive a combination of TPV 500mg/RTV 200 mg twice daily for 11 days (Days 3-13).
  On Day 12, subjects will receive a single 10 mg dose of rosuvastatin co-administered with TPV/r..
  Other Names: Crestor

SUMMARY:
Tipranavir (TPV) plus ritonavir (RTV) is indicated for use as part of an antiretroviral treatment regimen for resistant HIV-1 infection in adult patients. Since significant cholesterol and triglyceride elevations are commonly reported during TPV/RTV treatment, effective treatment strategies are critical to prevent long-term cardiovascular events. Rosuvastatin, a potent 3-hydroxy-3-methylglutaryl-coenzyme (HMG-CoA) reductase inhibitor, is unlikely to interact with TPV/RTV since it is not extensively metabolized, however, a formal drug interaction study is needed before this combination can be recommended. This study will examine the pharmacokinetic interactions between tipranavir/ritonavir (TPV/RTV [TPV/r] 500 mg/200 mg twice daily [B.I.D]) and single dose rosuvastatin when the two are co-administered to healthy adult volunteers. The investigators hypothesize that if tipranavir 500 mg is co-administered with low-dose ritonavir 200 mg and rosuvastatin (10 mg) no significant clinical interaction will occur.

DETAILED DESCRIPTION:
This is a prospective, open-label pharmacokinetic study in healthy HIV seronegative adults. This study will examine the pharmacokinetic interactions between steady-state TPV/r 500 mg/200 mg B.I.D. and single dose rosuvastatin 10 mg when the drugs are co-administered.

Rosuvastatin 24 hour pharmacokinetic sampling will be performed on days 1-2 and 12-13. Rosuvastatin 48 hr samples will be collected on days 3 and day 14.

Tipranavir and ritonavir 12 hour pharmacokinetic sampling will be on day 11 and 12.

Safety assessments (physical examination, vital sign measurements, and clinical laboratory tests) will be performed at screening, during the study and prior to discharge. Subjects will be continuously monitored for adverse events throughout the duration of the study.

On Day 1, subjects will receive a single 10 mg dose of rosuvastatin. Beginning on Day 3, subjects will receive a combination of TPV 500 mg/RTV 200 mg twice daily for 11 days (Days 3-13).

On Day 12, subjects will receive a single 10 mg dose of rosuvastatin co-administered with TPV/r.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a body mass index (BMI) of 18 to 30 kg/m2, inclusive (BMI = weight (kg)/[height (m)]2) and weigh at least 50 kg.
* Males or females, ages > 18 to < 65 years.
* Women of childbearing potential (WOCBP) must not be nursing or pregnant. All women of childbearing potential (have not reached menopause nor undergone hysterectomy, bilateral oophorectomy, or tubal ligation) must have a negative serum human chorionic gonadotropin (HCG) test performed at screening (within 24 hours before the start of study day 1). Female subjects who are not of reproductive potential (have reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) or whose male partner has undergone successful vasectomy with resultant azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Documentation of menopause, sterilization (hysterectomy, oophorectomy, tubal ligation, or vasectomy) and azoospermia by patient-reported history is acceptable. Both male and female study volunteers of reproductive potential must agree not to participate in a conception process (i.e., active attempt to become pregnant or to impregnate via sperm donation or in vitro fertilization), and, if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use a form of contraception as specified below while receiving protocol-specified medication(s) and for one month after stopping the medication(s). Male study volunteers will be required to use a barrier method for at least 3 months after completion of the study.

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide

Exclusion Criteria:

* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* History of acute or chronic pancreatitis.
* History of diabetes mellitus, hypertriglyceridemia, or chronic renal insufficiency.
* Proven or suspected acute hepatitis at the time of study entry.
* Current or recent (within 3 months) gastrointestinal disease which would interfere with the conduct or interpretation of the study.
* Any major surgery within 4 weeks of enrollment. Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of enrollment.
* Inability to tolerate oral medication.
* Inability to tolerate venipuncture and/or absence of secure venous access.
* Known or suspected HIV infection or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Known active drug or alcohol abuse which, in the opinion of the investigator, makes study participation to completion unlikely.
* Any other sound medical, psychiatric, and/or social reason, as determined by the investigator.
* Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin above the upper limit of normal.
* Hemoglobin < 9.5 g/dL, and platelet count < 100,000/mm3.
* Subjects with creatine phosphokinase (CPK) elevation greater than 3 times the upper limit of normal.
* Any other clinically significant screening lab abnormality (as determined by the investigator)
* History of any significant drug allergy, drug rash, or sensitivity to any class of drugs relevant to the study drugs.
* Prior exposure to tipranavir/ritonavir.
* Exposure to any investigational drug within 4 weeks of enrollment and throughout the study.
* Any previous hypersensitivity or intolerance to tipranavir or ritonavir or any other ingredient of Aptivus or Norvir.
* Hypersensitivity to sulfonamides
* Any previous hypersensitivity or intolerance to rosuvastatin or any other ingredient of Crestor (rosuvastatin).
* Known elevated liver enzymes in past clinical trials with any compound
* Use of any agent, within 2 weeks of dosing, that is known to induce or inhibit drug metabolizing enzymes
* Use of any over-the-counter drugs, including antacids, alternative herbal products, or prescription drugs that, in the opinion of the investigator, might interfere with the absorption, distribution, or metabolism of TPV, RTV, or rosuvastatin within 14 days of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To compare single dose rosuvastatin Area Under the Curve during 24 hours (AUC0-24h) and Cmax with single dose rosuvastatin AUC0-24h and Cmax when co-administered with TPV/r 500 mg/200 mg twice daily at steady state | 24 hours

SECONDARY OUTCOMES:
To evaluate the short term safety and tolerance of TPV/r (500 mg/200 mg B.I.D) combined with single dose rosuvastatin (10 mg) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pham, PharmD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a prospective, open-label pharmacokinetic study